CLINICAL TRIAL: NCT05384392
Title: Biomarkers Predictive of Thymic Evolution and Therapeutic Response at 2 Years in Patients With a First Psychotic Episode
Acronym: PEPAMARKER
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 29BRC21.0196
Record Dates: First submitted 2022-04-28; First posted 2022-05-20 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: First-episode Psychosis
Keywords: Bipolar Disorder; Schizophrenia
MeSH Terms: conditions — Bipolar Disorder; Schizophrenia | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Intervention (Experimental): All patients included in the study will be required to complete the examinations specified in the protocol.
  Interventions: Other: Recorded interview; Other: Clinical scales; Biological: Blood sample

INTERVENTIONS:
Other: Recorded interview — A recorded clinical interview, transcribed verbatim and blinded analyzed
Other: Clinical scales — Answering to clinical scales : PANSS (Positive and Negative Syndrome Scale); BPRS (Brief Psychiatric Rating Scale); CDSS (Calgary Depression Scale for Schizophrenia); MADRS (Montgomery-Åsberg Depression Rating Scale); Altman; YMRS (Young Mania Rating Scale); GAF (Global Assessment of Functioning); SF-36 (36-Item Short Form Survey); CGI-S (Clinical Global Impression Scale) et CGI-I (CGI-Improvement)
Biological: Blood sample — Blood collection of inflammatory markers (IL-1, sIL-2R, IL-4, IL-6, IL-8 and TNF levels) and 2 EDTA tubes and 2 dry tubes for biological collection (plasma bank and serum bank). This blood sample will be taken during routine sampling.

SUMMARY:
Psychosis is a severe, common, and disabling psychological disorder. An epidemiological study conducted in England reported an incidence of 34 new cases per 100,000 person-years, with a peak between 16 and 19 years of age. Following a first psychotic episode, two clinical evolutions are possible: thymic psychosis (17%) and non thymic psychosis (83%). The first includes bipolar disorders with a psychotic component and major depressive disorders with a psychotic component; the second, other psychotic disorders, mainly schizophrenia. One of the major difficulties encountered is the frequent impossibility of specifying the type of psychosis at the beginning of the psychotic episode. However, these disorders require different therapies, particularly medication. This leads to a delay in diagnosis with a high risk of relapse.

The semiological study of these diseases being carried out within the framework of interviews, it seems interesting to be able to record these and to obtain a quantitative and objective measurement through the study of language. The use of machine learning has made it possible to distinguish patients with schizophrenia from those with bipolar disorder by graphical analysis of language in a more efficient way than with clinical scales.Moreover, it is possible to identify linguistic markers: thus, an alteration of syntactic structures and prosody would be more present in non-thymic than in thymic psychoses.

Paraclinical markers are also emerging. In particular, the link between inflammation and mental disorders.For example, an increase in IL-8 has been found only in thymic psychoses.

In this context, it seems essential to be able to distinguish these disorders as early as possible through the combined use of clinical and paraclinical markers, and to be able to better understand their pathophysiology.

ELIGIBILITY:
Inclusion Criteria:

* Patient with a first episode of psychosis,
* Aged between 15 and 30 years,
* Able to consent and having signed a consent form (parental consent for minors).

Exclusion Criteria:

* Introduction or increase of antipsychotic and/or antidepressant and/or thymoregulatory treatment in the last month,
* Mother tongue other than French,
* Psychotic episode due to an organic disorder,
* Psychotic episode induced by the use or withdrawal of toxic substances with severe dependence ,
* Intellectual deficit,
* Chronic inflammatory disease,
* Immunomodulatory treatment,
* Contraindication to MRI,
* Pregnant or breastfeeding woman,
* Patient under court protection, guardianship, curatorship or deprived of liberty.

Ages: 15 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 217 (Estimated)
Dates: Start 2025-03-27 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2030-03 (Estimated)

PRIMARY OUTCOMES:
Evaluation of thymic evolution | Day 0, Year 2
  The primary endpoint is the thymic evolution (yes or no) of the initial psychotic episode The prosodic linguistic markers (fundamental frequency and latency) will be measured at Day 0 during a routine clinical interview and wil enable to build a predictive model to predict the thymic evolution at 2 years in patients with a first psychotic episode. This is main objective of study.
  The assessment will be measured the answer yes or no, at 2 years, at question, is the psychotic episode a thymic disorder?".

SECONDARY OUTCOMES:
Evaluation of thymic evolution according syntactic linguistic markers | Day 0
  The thymic evolution will be evaluated according syntactic linguistic markers at Day 0 during a clinical interview.
  Syntactic complexity is assessed using lexical density (%), lexical diversity (%), and the average number of words per clause. The use of the singular first-person pronoun "je" and speech disfluencies are also foregrounded in our project.
Evaluation of thymic evolution according semantic linguistic markers | Day 0
  The thymic evolution will be evaluated according semantic linguistic markers at Day 0 during a clinical interview.
  Semantic marker is grounded in a method for measuring semantic coherence called "latent semantic analysis (LSA)". LSA entails computing the cosine similarity between two vectors in each comparison of documents, i.e. between two sentences or between two turn-takings. Semantic coherence is consequently expressed by a value between -1 and 1.
Inflammatory markers | Day 0
  Assessment according inflammatory markers (IL-1, sIL-2R, IL-4, IL-6, IL-8 and TNF levels) at T0 during the initial biological work-up. The unit of measure is pg/mL for the inflammatory markers.
Evaluation of thymic evolution according PANSS | Day 0, Year 1, Year 2
  The thymic evolution will be evaluated according Positive and Negative Syndrome Scale (PANSS). The Positive and Negative Syndrome Scale (PANSS) is an established psychiatric rating system that is an operationalized, drug-sensitive instrument that offers balanced representation of positive and negative symptoms and estimates their relationship to one another and to global (or general) psychopathology. The scale has 30 items to explore and is scored from 1 (absence) to 7 (extreme).
Evaluation of thymic evolution according BPRS | Day 0, Year 1, Year 2
  The Brief Psychiatric Rating Scale (BPRS) is a tool clinicians or researchers use to measure psychiatric symptoms such as anxiety, depression, and psychoses.
  Persons having or suspected of having schizophrenia or other psychotic disorder manifest the disorder in multiple ways. The BPRS assesses the level of 18 symptom constructs such as hostility, suspiciousness, hallucination, and grandiosity. It is particularly useful in gauging the efficacy of treatment in patients who have moderate to severe psychoses.
  It is based on the clinician's interview with the patient. The rater enters a number for each symptom construct that ranges from 1 (not present) to 7 (extremely severe).
Evaluation of thymic evolution according CDSS | Day 0, Year 1, Year 2
  This scale is designed to assess depression in people with schizophrenia. The questionnaire consists of 9 items (depressed mood, hopelessness, self-deprecation, guilt-themed reference thoughts, pathological guilt, morning depression, early arousal, suicidal ideation, and observed depression) covering the last 2 weeks.
  4-point Likert-type scale ranging from 0= "absent" to 3= "severe" for each items. More higher score = More severe symptoms.
Evaluation of thymic evolution according MADRS | Day 0, Year 1, Year 2
  The Montgomery-Åsberg Depression Rating Scale (MADRS) is a scale used to assess the severity of depression in patients with mood disorders. It is also frequently used to measure changes brought about by treatment of depression.
  It assesses the severity of symptoms in a wide range of areas such as mood, sleep and appetite, physical and psychological fatigue and suicidal ideation.
  The scale has 10 items rated from 0 to 6 (> 34 points: the patient is considered to be in severe depression).
Evaluation of thymic evolution according Altman | Day 0, Year 1, Year 2
  The Altman Self-Rating Scale is a short 5-item self-report questionnaire that can be useful in assessing the presence and severity of manic or hypomanic symptoms.
  Each of these points has five statements that correspond to scores of 0 to 4; 0 being unchanged from "normal" or baseline, to 4 being clearly manic thoughts or behavior. The subject is asked to choose one statement from each of the five domains that best describes how they have felt over the past week.
  Scores above 5 indicate mania or hypomania, with the severity of symptoms increasing with higher scores.
  Because this scale is consistent with diagnostic criteria, it can be used effectively as a screening and diagnostic tool despite its brevity.
Evaluation of thymic evolution according YMRS | Day 0, Year 1, Year 2
  The Young Mania Rating Scale (YMRS) is one of the most frequently utilized rating scales to assess manic symptoms. The scale has 11 items and is based on the patient's subjective report of his or her clinical condition over the previous 48 hours.
  The YMRS total score ranges from 0 to 60 where higher scores indicate more severe mania.
Evaluation of thymic evolution according GAF | Day 0, Year 1, Year 2
  The Global Assessment of Functioning, or GAF, scale is used to rate how serious a mental illness may be. It measures how much a person's symptoms affect their day-to-day life on a scale of 0 (minimum value) to 100 (maximum value). It's designed to help mental health providers understand how well the person can do everyday activities. The higher subject score, the better subject is able to handle daily activities.
Evaluation of thymic evolution according SF-36 | Day 0, Year 1, Year 2
  SF-36 is a set of generic, coherent, and easily administered quality-of-life measures. These measures rely upon patient self-reporting and are now widely utilized for routine monitoring and assessment of care outcomes in adult patients.
  The SF-36, as described in the name, is a 36-item patient-reported questionnaire that covers eight health domains: physical functioning (10 items), bodily pain (2 items), role limitations due to physical health problems (4 items), role limitations due to personal or emotional problems (4 items), emotional well-being (5 items), social functioning (2 items), energy/fatigue (4 items), and general health perceptions (5 items). Scores for each domain range from 0 to 100, with a higher score defining a more favorable health state.
Evaluation of thymic evolution according CGI | Day 0, Year 1, Year 2
  Amongst the most widely used of extant brief assessment tools in psychiatry, the CGI is a scale that measures illness severity (CGIS) and global improvement or change (CGIC). The illness severity and improvement sections of the instrument are used frequently in both clinical and research settings. This scale asks that the clinician rate the patient relative to their past experience with other patients with the same diagnosis, with or without collateral information. The CGI has proved to be a robust measure of efficacy in many clinical drug trials, and is asy and quick to administer, provided that the clinician knows the patient well.
  The CGI is rated on a 7-point scale, with the severity of illness scale using a range of responses from 1 (normal) through to 7 (amongst the most severely ill patients). CGI-C scores range from 1 (very much improved) through to 7 (very much worse). Each component of the CGI is rated separately; the instrument does not yield a global score.

CONTACTS AND LOCATIONS:
Locations (6):
- France (6):
  - Dr Bénédicte GOHIER, Angers
  - Dr Florian STEPHAN, Brest
  - Dr Anne SAUVAGET, Nantes
  - Dr Sonia MARSELLA, Quimper
  - Dr Dominique DRAPIER, Rennes
  - Dr Vincent CAMUS, Tours

IPD SHARING:
Plan to Share IPD: Yes
All collected data that underlie results in a publication
Supporting Information: Study Protocol
Time Frame: Data will be available after the publication of result and ending fifteen years following the last visit of the last patient.
Access Criteria: Data access requests will be reviewed by the internal committee of BrestUH. Requestors will be required to sign and complete a data access agreement.

REFERENCES:
- [Derived] Terrisse R, Lemey C, Kim-Dufor DH, Miglianico L, Stephan F. PEPAMARKER: a multicenter cohort study protocol on predictive biomarkers of affective vs. non-affective trajectories in first-episode psychosis. Front Psychiatry. 2026 Jan 14;16:1702187. doi: 10.3389/fpsyt.2025.1702187. eCollection 2025. PMID 41614097